CLINICAL TRIAL: NCT01047059
Title: Clinical Pilot to Evaluate the Accuracy of FDG-/FLT-PET and DCE-MRI for Early Prediction of Non-Progression in Patients With Advanced Non Squamous Cell Non Small Cell Lung Cancer (NSCLC) Treated With Erlotinib and Bevacizumab and to Associate Imaging Findings With Molecular Markers
Brief Title: Molecular Imaging With Erlotinib and Bevacizumab
Acronym: MIMEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Prof. Dr., Lung Cancer Group Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIMEB; 2009-012607-26 (EudraCT Number)
Record Dates: First submitted 2010-01-10; First posted 2010-01-12 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trial Intervention (Experimental): 150mg Erlotinib daily, 15mg/kg b.w. Bevacizumab on d1, d22, d43 as medication FDG-PET, FLT-PET and DCE-MRI as diagnostical tools
  Interventions: Drug: Erlotinib, Bevacizumab; Drug: Fluoro-D-glucose; Drug: Fluoro-L-thymidine; Drug: Gadolinium-DPTA

INTERVENTIONS:
Drug: Erlotinib, Bevacizumab — Erlotinib 150mg/d d1-d43 p.o. Bevacizumab 15mg/kg b. w. d1, d22, d43 i.v.
  Other Names: Tarceva; Avastin
Drug: Fluoro-D-glucose — Tracer for PET imaging
  Other Names: FDG-PET
Drug: Fluoro-L-thymidine — FLT-PET tracer for imaging
  Other Names: FLT-PET
Drug: Gadolinium-DPTA — Contrast agent for DCE-MRI imaging
  Other Names: Gd-DPTA; Magnevist

SUMMARY:
The patients will be treated with erlotinib and bevacizumab for a six-week period. Imaging procedures will be performed at baseline, after one week of therapy and after the six weeks of treatment.

The combination of erlotinib and bevacizumab represents an effective therapeutic strategy in NSCLC with the highest response rates ever reported for relapsed NSCLC having been observed recently in a phase II trial. Early differentiation of patients profiting and of patients not profiting from this therapy is of major relevance for further improving this targeted therapy approach and to develop more effective, personalized treatment strategies. We aim at this early identification by the combination of molecular and functional imaging tools (FDG-, FLT-PET, DCE-MRI), molecular marker analyses in tissue and peripheral blood (EGFR- and KRAS mutational status and high throughput mutational profiling in tumor tissue, angiogenesis-associated biomarkers and expression profiling in peripheral blood) and pharmokokinetic analyses. From the combined analyses of these tools we expect a better understanding of the host-drug interaction as a precondition for further improvement of erlotinib-bevacizumab combination therapy in NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven non-squamos NSCLC stage IIIB with pleural effusion or stage IV
* ≥ 18 years of age
* Performance status ECOG 0-2
* Estimated life expectancy of at least 12 weeks
* Subjects with at least one measurable or nonmeasurable (CT or MRI) lesion according to RECIST
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1,500 /mm3
* Platelet count ≥ 100 000/μL
* Total bilirubin ≤ 2 x ULN
* ALT, AST and alkaline phosphatase (AP) ≤ 2,5 x ULN
* PT-INR/PTT < 1.5 x ULN
* Creatinine clearance (CrCl) ≥ 60 ml/min calculated by either Cockcroft-Gault or by 24 hours urine collection
* Written informed consent (after adequate explanation of the trial) to participate in the trial and to adhere to trial procedures, as well as consenting to data protection procedures
* No clinical or radiological sign of interstitial lung disease, no interstitial lung disease in the past
* Patients must be able to take oral medication
* In case of female patients with childbearing potential:
* negative serum or urine HCG in women with childbearing potential
* effective method of contraception (Pearl-Index not greater than 1%)
* at least 12 months after last menstruation

Exclusion Criteria:

* Patient has received prior chemotherapeutic regimens for advanced disease. Prior chemotherapy given as neoadjuvant or adjuvant therapy for early stage disease, completed at least 12 months prior to diagnosis of advanced stage disease, will not be considered as exclusion criterion.
* Patient has received prior EGFR-targeted therapy
* Squamous-cell carcinoma (SCC) histology, SCLC histology or mixed histology
* Evidence of tumor invading or abutting major blood vessels
* Patient has signs or symptoms of acute infection requiring systemic therapy (acute or within the last 14 days)
* Uncontrolled diabetes mellitus with HbA1c > 7,5% or elevated blood glucose levels levels of > 200 mg/dL
* History of uncontrolled heart disease (congestive heart failure > NYHA class 2; active Coronary Arterial Disease (CAD), (MI more than 6 months prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (except, when controlled by beta blockers or digoxin) and/or uncontrolled hypertension (> 150/100 mmHg)
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of erlotinib and (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection, total parenteral nutrition with lipids)
* History of HIV infection or previously sero-positive for the virus
* History of Hepatitis B or/and C or previously sero-positive for the Hepatitis B or/and C virus
* Patients with seizure disorder requiring CYP3A4-inducing anti-epileptics
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* History of thrombotic disorders within the last 6 months prior to enrolment
* Fine needle biopsy or open biopsy within 1 week prior inclusion
* Clinically symptomatic leptomeningeal or brain metastases (patients with clinically stable brain metastases may be enrolled)
* Impaired wound healing, non-healing wounds, ulcers, fractures or any condition that provokes uncontrolled bleeding
* Preexisting neuropathia ≥ grade 2 • History of grade ≥2 hemoptysis (bright red blood of at least 2.5 ml)
* Patients undergoing renal dialysis
* Past or current history of cancer other than the entry diagnosis EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* Any person being in an institution on assignment of the respective authority
* Urine protein qualitative value of > 30 in urinalysis or > +1 in proteinuria testing by dipstick
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
* Concomitant or intented anticoagulation therapy
* Planned surgical or dental invasive intervention (e.g. tooth extraction, planned surgeries) during the course of the study
* Any serious medical condition with organ impairment
* Hypersensitivity to bevacizumab or erlotinib or any of their ingredients
* Major surgery or significant traumatic injury within the last 4 weeks before inclusion
* Parallel participation in another clinical trial or participation in another clinical trial within the last 30 days or 7 half-life's, whatever is of longer duration, prior study start
* Pregnancy, breast feeding
* Claustrophobia
* Known allergic reaction to Gadolinium
* Heart pacemaker
* Ferromagnetic and electronic implants in special locations (e. g. cerebral)
* Cochlea implants
* known allergic reaction to non-ionic iodinated computed tomography contrast agents
* known hyperthyroidism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of imaging findings in FDG-/FLT-PET and DCE-MRI after one week of treatment for early prediction of RECIST-based non-progression and progression-free survival after 6 weeks of therapy | 24 months

SECONDARY OUTCOMES:
Correlation of mutational profiling with imaging characteristics Prognostic accuracy of imaging Pharmacokinetic analysis Reliability of DCE-MRI Correlation of peripheral biomarkers with clinical outcome, mutational profiling, imaging characteristics | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wolf, MD, Prof., Principal Investigator — Lung Cancer Group Cologne (LCGC); Matthias Scheffler, MD, Study Chair — Lung Cancer Group Cologne (LCGC); Lucia Nogova, MD, Study Chair — Lung Cancer Group Cologne (LCGC)
Locations (1):
- Center for Integrated Oncology (CIO), University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany